CLINICAL TRIAL: NCT04945109
Title: The Effect of Wolffia Globosa (Mankai) on Glycemic Control Among Patients With Type 2 Diabetes; A Randomized Crossover Controlled Trial
Brief Title: Wolffia Globosa (Mankai) and Glycemic Control Among Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Iris Shai, Prof. Iris Shai, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0094-21SOR
Record Dates: First submitted 2021-06-14; First posted 2021-06-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Water

STUDY DESIGN:
Intervention Model Description: A randomized cross-over, 4-week trial, where participants will be allocated to start with or without daily Mankai supplementation (fresh Mankai beverage) added on top of a standardized diabetes-related healthy diet, each for two weeks. The investigators will follow postprandial and overnight glycemic response using ﬂash glucose monitoring system device. Other outcomes include clinical parameters (weight, waist circumference, blood pressure), blood, urine, fecal measurements, overall appetite/ satiety, food intake consumption, symptoms, and medical treatment.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mankai beverage first (Experimental): Two weeks of Mankai supplementation followed by two weeks of water supplement
  Interventions: Other: Mankai beverage; Other: Water (control)
- Mankai beverage last (Experimental): Two weeks of water supplementation followed by two weeks of Mankai supplement
  Interventions: Other: Mankai beverage; Other: Water (control)

INTERVENTIONS:
Other: Mankai beverage — Recommended background healthy diet with Mankai supplementation after main meal (300 ml)
Other: Water (control) — Recommended background healthy diet with water supplementation after main meal (300 ml)

SUMMARY:
The investigators primarily aim to explore the effect of daily additive supplementation of Mankai on glucose control among participants with T2D.

DETAILED DESCRIPTION:
Type 2 diabetes is a major public health concern in Western societies. Type 2 diabetes is associated with high morbidity and shorter life expectancy. In patients with type 2 diabetes maintaining glycemic control is associated with lower rates of complications and mortality associated with the disease. Thus, there is a great need to recognize nutritional elements that improve glycemic control and insulin sensitivity in patients with type 2 diabetes. Mankai, a strain of Wolffia globosa recently developed under controlled conditions, is characterized by high protein content and good bioavailability of proteins, rich in soluble fiber, vitamins (including vitamin B12), minerals (including iron and zinc), omega 3 fatty acids, and polyphenols. The 18-month long DIRECT PLUS trial was a weight-loss intervention conducted among 294 participants with abdominal obesity or dyslipidemia. 98 of the study participants were assigned to the intervention of a green Mediterranean diet and were instructed to consume four frozen cubes of Mankai daily. Main conclusions from the DIRECT PLUS refer to the beneficial effect of the green-Mediterranean diet on cardiometabolic risk, gut bacteria, and liver fat, with no evidence of disadvantages or adverse effects of long-term Mankai consumption. In 2019, the investigators reported that among non-diabetics and those with fasting glucose levels within the normal range, consuming a Mankai smoothie in the evening led to lower glucose levels after the meal and lower fasting overnight compared to a yogurt smoothie. The investigators now plan to explore the effect of Mankai daily supplementation on post-meal glycemic response in participants with type 2 diabetes. The investigators hypothesize that the addition of Mankai consumption after a meal may mitigate glucose excursions compared with control.

ELIGIBILITY:
Inclusion Criteria:

* Age => 30 years
* A formal diagnosis of T2D (126mg/dl fasting glucose or higher, or HbA1c=>6.5%) or taking T2D medications.

Exclusion Criteria:

* Treatment with coumadin (warfarin)
* Advanced renal failure
* A significant illness that might require hospitalization
* State of pregnancy or lactation
* Presence of active cancer or chemotherapy treatment in last three years
* Participation in another trial.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Changes in glycemic control | Through study completion, 24hours a day (continuous measurement, all day, 4 weeks)
  Continuous glucose excursions monitoring

SECONDARY OUTCOMES:
Insulin | 0, 2, 4 weeks
  Blood measured insulin (mIU/L)
Fasting glucose | 0, 2, 4 weeks
  Blood measure of glucose (mg/dL)
Serum lipids | 0, 2, 4 weeks
  Lipid profile: TC, TG, HDL, LDL
Serum liver Enzymes | 0, 2, 4 weeks
  Liver enzymes: ALT, AST, GGT, ALKP (U/l)
Inflammation | 0, 2, 4 weeks
  hs-CRP
Microbiota profile | 0, 2, 4 weeks
  Fecal bacterial composition and richness
CBC | 0, 2, 4 weeks
  Complete blood cells count: red, white, differential
Anthropometric | 0, 2, 4 weeks
  Weight (kg), height (cm) to calculate BMI (kg/m^2)
Abdominal obesity | 0, 2, 4 weeks
  Waist circumference (cm)
Pulse | 0, 2, 4 weeks
  Resting pulse (beats per minute)
Blood pressure | 0, 2, 4 weeks
  Systolic and Diastolic blood pressure (mmHg)
Urine markers of glucose | 0,2,4 weeks
  Glucose in urine (mmol/L)
Urine markers of protein | 0,2,4 weeks
  Protein in urine (mg/day)
questionnaire 1 | 0, 2, 4 weeks
  Self reports on symptoms during the intervention (yes/no questions)
questionnaire 2 | 0, 2, 4 weeks
  Self reports on appetite during the intervention (scale of 0-100%)
questionnaire 3 | 0, 2, 4 weeks
  Self reports on satiety during the intervention (scale of 0-100%)
questionnaire 4 | 0, 2, 4 weeks
  Self reports on lifestyle (daily log, self report without scale of measurement)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Tirosh, MD PhD, Principal Investigator — Sheba Medical Center
Locations (2):
- Israel (2):
  - Nuclear research center Negev, Dimona
  - Sheba Medical Centre, Ramat Gan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zelicha H, Kaplan A, Yaskolka Meir A, Tsaban G, Rinott E, Shelef I, Tirosh A, Brikner D, Pupkin E, Qi L, Thiery J, Stumvoll M, Kloting N, von Bergen M, Ceglarek U, Bluher M, Stampfer MJ, Shai I. The Effect of Wolffia globosa Mankai, a Green Aquatic Plant, on Postprandial Glycemic Response: A Randomized Crossover Controlled Trial. Diabetes Care. 2019 Jul;42(7):1162-1169. doi: 10.2337/dc18-2319. Epub 2019 May 10. PMID 31076421